CLINICAL TRIAL: NCT06802042
Title: Effect of Lactobacillus DSM17938+ on Functional Constipation and Intestinal Flora in Pregnant Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K6993
Record Dates: First submitted 2025-01-25; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Functional Constipation (FC)
MeSH Terms: interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group (Experimental): The intervention group (n=20) received free intervention with probiotic bacteria (Lactobacillus reuteri DSM17938+) for 4 weeks (1 bag bid)
  Interventions: Other: Intervention with probiotic bacteria
- control group (Active Comparator): The control group (n=20) received lactulose oral solution free of charge for 4 weeks (1-2 bags qd for the first three days, and then increased or reduced according to constipation)
  Interventions: Drug: Lactulose oral solution treatment

INTERVENTIONS:
Other: Intervention with probiotic bacteria — The intervention group (n=20) received free intervention with probiotic bacteria (Lactobacillus reuteri DSM 8 +) for 4 weeks (1 bag bid)
  Arms: intervention group
Drug: Lactulose oral solution treatment — The control group (n=20) received lactulose oral solution free of charge for 4 weeks (1-2 bags qd for the first three days, and then increased or reduced according to constipation)
  Arms: control group

SUMMARY:
Constipation (constipation) is a common clinical symptom, including difficulty in defecation and / or reduced frequency of defecation, dry and hard stool, difficulty in defecation, feeling of inexhaustible defecation, feeling of anorectal obstruction, time-consuming defecation and need for auxiliary defecation. Reduced defecation means defecation less than 3 times a week.Constipation is very common during pregnancy, and studies have found that the incidence of constipation in pregnant women is as high as 40%. Among them, the prevalence of functional constipation in the early, middle, late and postpartum pregnancies is 35%, 39%, 21% and 17% respectively, with the highest in the early and middle pregnancies.Constipation can increase the psychological burden of pregnant women and affect their quality of life. Long-term severe constipation can also induce or aggravate hemorrhoids. Severe constipation can induce uterine contractions, which will adversely affect the pregnancy outcome of pregnant women.Studies have found that there is a difference in the abundance of intestinal flora between patients with constipation during pregnancy and pregnant women without digestive tract diseases.Although microecological preparations are not front-line drugs for the treatment of chronic constipation, they can promote intestinal peristalsis and the recovery of gastrointestinal motility by regulating the imbalance of intestinal flora. More and more researchers recommend them as long-term adjuvant drugs for chronic constipation. Probiotics are a type of microecological preparation, which refers to living microorganisms that can have beneficial health effects on the host after ingesting a sufficient amount.It is relatively safe to supplement probiotics during pregnancy.Our research team found a probiotic strain, Lactobacillus reuteri DSM17938+, which has no significant difference in improving constipation symptoms in patients with constipation compared with lactulose, and is even more effective than lactulose in alleviating abdominal pain and flatulence symptoms.However, clinical studies proving that Lactobacillus reuteri DSM17938 + is effective on constipation are generally concentrated abroad, and mainly focus on infants and young children, children, adults] or intestinal colic. Data on maternal population in China is lacking.

ELIGIBILITY:
Inclusion Criteria:

* (1) Pregnant women, age ≥18 years and <40 years old, and gestational age <28 weeks; (2) Must meet two or more of the following symptoms (Refer to the Roman IV standard):

  * It is difficult to defecate at least 25% of the time;

    * It is lumpy or hard stool at least 25% of the time;

      * It is not enough to defecate at least 25% of the time;

        * It is at least 25% of the time that there is anorectal obstruction or obstruction in defecation;

          * It requires manual assistance at least 25% of the time;

            ⑥It is spontaneous defecation less than 3 times a week. At the same time, loose stools rarely occur when no laxatives are used, which does not meet the diagnostic criteria of irritable bowel syndrome (IBS). The symptoms in the past 2 weeks have met the above diagnostic criteria.

            (3) Pregnant women receive and follow high-protein and high-fiber dietary guidance during the first trimester.

            (4) There were no other complications. (5) No medication was used to interfere with constipation symptoms.

Exclusion Criteria:

* (1) Non-pregnant women, age <18 years or ≥40 years old, and gestational age ≥28 weeks; (2) Constipation caused by intestinal and systemic organic factors, drugs and other reasons, or concurrent with other non-constipation intestinal diseases; (3) History of use of antibiotics, probiotics, prebiotics, etc. in the past 2 weeks; (4) Pregnant women with thyroid disease, diabetes, hypertension, obesity, overweight or any metabolic disease.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of probiotic bacteria (Lactobacillus reuteri DSM17938+) on functional constipation in pregnant women during the first and second trimester | From enrollment to the end of treatment at 4 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Chinese Academy of Medical Science & Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Wenzhou People's Hospital, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No